CLINICAL TRIAL: NCT01979575
Title: An Observational Study on the Effects of Steep Trendelenburg Position and Pneumoperitoneum on Hemodynamic Changes Observed With Non-invasive Cardiac Monitors
Brief Title: Trendelenburg Study
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 495567
Record Dates: First submitted 2013-11-01; First posted 2013-11-08 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Comparison of Non-invasive Monitors of Cardiac Function
Keywords: Nexfin; Flotrac; Esophageal; Cardiac output

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
1) Observe the hemodynamic and cardiovascular changes associated with the change from the supine to the steep Trendelenburg position, 2) Observe the hemodynamic and cardiovascular changes during intra-abdominal insufflation used during laparoscopic surgical procedures.

DETAILED DESCRIPTION:
This is a single site, prospective, non-blinded, non-randomized, non-interventional study designed to evaluate the hemodynamic and cardiovascular effects of the steep Trendelenburg position on non-invasive or minimally invasive monitors used in the operating room during surgical procedures requiring this patient position.

SPECIFIC AIMS: 1) Observe the hemodynamic and cardiovascular changes associated with the change from the supine to the steep Trendelenburg position. 2) Observe the hemodynamic and cardiovascular changes during intra-abdominal insufflation used during laparoscopic surgical procedures.

HYPOTHESIS: Hemodynamic and cardiovascular changes during alterations in position from supine to steep Trendelenburg and intra-abdominal insufflation measured by non-invasive and minimally invasive monitors will correlate with transthoracic echocardiographic measurements.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective surgery requiring steep trendelenburg positioning.

Exclusion Criteria:

* BMI >30. <18 years. Pregnancy. Prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective surgery.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
An observational study on the effects of steep Trendelenburg position and pneumoperitoneum on hemodynamic changes observed with non-invasive cardiac monitors | One year.
  Changes in cardiac output associated with patient position.

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Health System, Sacramento, California, United States